CLINICAL TRIAL: NCT06230081
Title: Postoperative Analgesia in Patients Undergoing Hip and Knee Replacement Surgery - a Study Comparing Ultrasound-guided Nerve Blocks With Intraoperative Local Anesthetic Infiltration or Opioids
Brief Title: Comparison Between Blocks or Not in Joint Arthroplasty
Acronym: BLAST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLAST study
Record Dates: First submitted 2024-01-04; First posted 2024-01-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis of the Knee or Hip
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Clonidine

STUDY DESIGN:
Intervention Model Description: The patients are randomized to either block or no block therapy
Who Masked: Outcomes Assessor
Masking Description: Nurses and physiotherapists evaluating the patients are blinded as well as the physician compiling the data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block (Active Comparator): Hip Arthroplasty: Multimodal analgesic therapy + Ultrasound guided PENG block and Iliohypogastric block or LFCN-block.
  Knee arthroplasty: Multimodal analgesic therapy + Ultrasound guided iPACK block, triple Genicular blocks, Vastus intermedius block, Adductor canal block and AFCN-block.
  Interventions: Drug: Ropivacain 5 mg/ml + Clonidine
- No block (No Intervention): Hip Arthroplasty: Multimodal analgesic therapy
  Knee Arthroplasty: Multimodal analgesic therapy + LIA

INTERVENTIONS:
Drug: Ropivacain 5 mg/ml + Clonidine — Drug used in the block
  Arms: Block

SUMMARY:
The purpose of this study is to evaluate the effect on postoperative pain, opioid consumption and function by adding a combination of regional blocks with local anaesthetic before total hip- and knee arthroplasty compared to standard pain management strategies.

DETAILED DESCRIPTION:
400 patients with osteoarthritis of the knee (200) or hip (200) necessitating total hip- or knee replacement are entered into the study. All patients are given a standard protocol of analgesics pre- and postoperatively. Patients are receiving general- or spinal anaesthesia during the surgery. General anaesthesia is conducted using Remifentanil 50ug/ml and Propofol 20 mg/ml utilizing a TCI protocol. The airway is managed by LMA or endotracheal tube. Spinal anaesthesia is conducted using isobaric Bupivacaine (hip) and hyperbaric bupivacaine (knee). Decision regarding type of anaesthesia is following guidelines of our department taking contraindications and patients preference into account.

Patients randomized to the block-group undergoing hip replacement surgery with posterior approach are given och combination of PENG block and Iliohypogastric block using Ropivacain 5 mg/ml with a total dose of 200 mg along with clonidine in a total dose of 75 micrograms. Patients undergoing hip replacement with lateral approach are given a combination of PENG block and LFCN block using Ropivacain 5 mg/ml with a total dose of 125 mg along with clonidine in a total dose of 56,25 micrograms. Patients randomized to the standard pain management strategy undergoing hip replacement surgery are given a combination of opioids, paracetamol and Cox-II inhibitors.

Patients randomized to the block-group undergoing knee replacement surgery are given a combination of iPACK-, genicular-, AFCN-, adductor canal and vastus intermedius block using Ropivacain 5 mg/ml with a total dose of 225 mg along with clonidine in a total dose of 75 micrograms. Patients randomized to the standard pain management strategy undergoing knee replacement surgery are given a perioperative periarticular LIA using Ropivacaine 300 mg along with 0,5 mg of adrenaline.

The randomization is executed on the day before surgery by opening of a closed numbered envelope giving information if the specific patient should have a block (intervention) or not (control). There are 200 prepared envelopes for the hip replacements and 200 for the knee replacements, with 100 blocks and 100 no blocks for each type. The envelopes are prepared by block randomization performed by computer software. Nurses and physiotherapists who evaluate postoperative pain are blinded from the intervention. The physician compiling the data from the study is also blinded to the intervention.

Preoperatively, information is collected regarding doses of analgesics and pain in everyday life is evaluated using the NRS scale. Preoperative pain is evaluated at rest and during mobilization.

Postoperatively, an evaluation of pain is made. After the operation the patients are monitored at the ward by the nurses and physiotherapists. The registration takes place using the subjective Numeric Rating Scale (NRS) and the objective Critical-Care Pain Observation Tool (CPOT). Pain is continuously evaluated during the hospital stay. The final registration takes place at the return visit 14 days after surgery. During the hospital stay, other parameters such as opioid consumption, requirement for urinary catheter, postoperative nausea and vomiting (PONV), time to mobilization and neurological complications are also registered. The number of extra opioid doses the patient requires are also registered. The number of days the patients need to stay in hospital after surgery are registered.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee- or hip necessitating total knee- or hip replacement
* Patients who understand the conditions of the study and are willing to participate for the length of the prescribed follow-up

Exclusion Criteria:

* Known allergy to local anesthetics or other contraindication for the use of local anesthetics.
* Coagulopathy
* Bilateral operation
* Revision arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in Postoperative pain assessed by NRS | The day of surgery, postop day 1 and 14 days post-surgery
  Patient experienced postop pain assessed by NRS (0-10)

SECONDARY OUTCOMES:
Difference in analgesia consumption | The day of surgery, postop day 1 and 14 days post-surgery
  Difference in extra oral- and intravenous analgesia consumption (tablets or injections - in mg)
Time to mobilization | The day of surgery, postop day 1
  Difference in time mobilizing to standing after surgery
Incidence of postoperative nausea and vomiting | The day of surgery, postop day 1
  Difference in postoperative nausea and vomiting (reported frequency)
Difference in postoperative pain depending on method of anesthesia | The day of surgery, postop day 1 and 14 days post-surgery
  Difference in postoperative pain depending on method of anesthesia, i.e. General- or Spinal anesthesia. Assessed by NRS (0-10)
urine catheter usage | 1-5 days post-surgery
  Difference in frequency of urine catheter usage
neurological complications | The day of surgery, postop day 1 and 14 days post-surgery
  Difference in frequency of neurological complications (reported to and assessed by physiotherapist)
Days in hospital | 1-5 days post-surgery
  Number of postoperative days in hospital
opioid consumption 14 days | 14 days post-surgery
  Difference in opioid consumption 14 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Flivik, MD PhD, Principal Investigator — Department of Orthopedics, Skane Univ Hosp
Locations (1):
- Dept of Anaesthesiology, Trelleborg Hospital, Trelleborg, Sweden

IPD SHARING:
Plan to Share IPD: No
General unidentified data and study protocol are available on request